CLINICAL TRIAL: NCT02610686
Title: Evaluating the Efficacy of Chloroquine for the Treatment of Plasmodium Vivax Infections in Central Vietnam
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Malariology, Parasitology and Entomology, Vietnam (Other Government)
Collaborators: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITM- NIMPE
Record Dates: First submitted 2015-10-23; First posted 2015-11-20 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2015-10

CONDITIONS: Plasmodium Vivax
Keywords: Plasmodium vivax; recurrence; drug resistance
MeSH Terms: conditions — Malaria, Vivax; Recurrence | interventions — Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chloroquine (Other): Single treatment arm
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Chloroquine — efficacy of chloroquine for the treatment of Plasmodium vivax infections
  Other Names: Nivaquine

SUMMARY:
Understanding the extent and regional distribution of CQR vivax malaria and detecting early signs of resistance is critical to prevent the spread of resistant strains, optimize treatment guidelines, and reduce the risk of recurrent and severe malaria. In Vietnam, CQR in P.vivax has been reported sporadically. One study carried out in Binh Thuan province (central-south Vietnam) at the end of the 1990s demonstrated early P.vivax recurrences (7%) by Day 16 after a 3-day CQ treatment. However, in a summary report to World Health Organization (WHO) including data from 11 sentinel sites, from studies conducted between 2006 and 2011 in central and southern Vietnam (total 350 patients), P.vivax is still considered sensitive to CQ. More recently in a cohort study conducted in Quang Nam province (Central Vietnam) in which P.vivax patients were treated radically with CQ and primaquine (10-day at 0.5mg/kg/day) following national guidelines, the 28-day failure rate was measured at 3.45% and CQ blood concentrations measured at day of recurrence (>100ng/ml) confirmed resistance in three patients. The current national guidelines for the radical cure regimen of P.vivax infections recommends 3 days of CQ (total 25 mg/kg body weight (bw)) together with 14 days of primaquine at 0.25 mg/kg bw/ day.

The current WHO protocol recommends a 28-day follow-up to assess the efficacy of CQ for the treatment of P.vivax infections. However, recurrence of early stage resistant parasites may occur after Day 28 in the presence of CQ blood levels above the minimum efficacy concentration (MEC, ≥100ng/ml) and relapses could occur as early as 36 days after standard CQ treatment. Therefore, in order to confirm CQR it is recommended to extend the follow-up period, to Day 42 or 63 and measure whole blood CQ level at Day 28 and at the time of recurrence. Moreover, it has been shown that emerging drug resistance in P.vivax is associated with delayed parasite clearance after treatment, i.e. some parasites are still detectable at Day 3. The aim of the present study is to assess the in vivo and ex vivo susceptibility of P.vivax to CQ in Central Vietnam following the currently recommended radical cure regimen and using GMP certified CQ.

DETAILED DESCRIPTION:
3.1 Study Design This study is designed as a 42-day drug efficacy study to evaluate clinical and parasitological responses after treatment of P.vivax malaria infections. Symptomatic patients with P. vivax mono-infections, meeting the study criteria, will be enrolled into the study, and treated with CQ (total dose 25gm/kg over 3 days). The treatment will be directly observed and the patients will be actively followed-up for 42 days according to an extended WHO protocol. At the end of the follow-up time, all patients will be treated with primaquine following national guidelines for the radical cure of P.vivax infections.

3.2 Study Site and Population The study will be carried out in Krong Pa district, Gia Lai province where both P.falciparum and P.vivax malaria incidence are among the highest in the country. The study will be located in Chu'R Cam commune where the study team will be working with the local health staff and all surrounding communes with malaria patients.

The local population is mainly composed by the JaRai ethnic minority and the main occupation consist of slash and burn agriculture (mainly maize, manioc and rice) in forest fields, together with seasonal work in rubber plantations, and small-scale production of goods for daily subsistence or trade e.g. coffee and cashew nuts. The climate is tropical with the dry season from November to April and the rainy season from May to October. The area is hilly and forested (secondary forest) and the main malaria vector is Anopheles dirus.

3.4 Trial Population The target population includes all P.vivax infected patients (children and adults) either presenting spontaneously at the CHC or identified through active screening in the community.

3.5 Trial Procedures 3.5.1 Screening and recruitment All consulting patients who meet the basic enrolment criteria during screening will be assigned a consecutive screening number and evaluated in greater depth by the medical doctor. Once the patient meets all the enrolment criteria, he or she (or a parent or guardian in case of children) will be asked for consent to participate in the study. Then, he/she will be allocated a study number (ID=sequential numbering). Any person who decides not to participate in the study will be examined, treated and followed-up by the health facility staff according to the standard of care established by the Ministry of Health.

At enrolment (Day 0) the patient will be and examined and a standardized pre-coded questionnaire will be filled in. A venous blood sample will be collected into sterile vacutainer tubes containing EDTA or acid-citrate-dextrose (EDTA/ACD) from all patients at enrolment. A minimum of 5ml of blood -and maximum of 8 ml- will be collected from adults, and 1ml/kg up to 5ml will be collected from children. Two blood drops will be added into a 1.5 ml tube containing 500 µL of RNAprotect reagent (Qiagen).

3.5.2 Treatment All patients will receive a full treatment with CQ at a dose of 25 mg of CQ base per kg body weight (bw) given over 3 days and under direct supervision. Patients will be observed for 60 minutes after treatment for adverse reactions or vomiting. Those patients vomiting their medication within the first 30 minutes will receive a repeat full dose; those vomiting from 30-60 minutes will receive half dose. If the patient vomits again, he or she will be withdrawn and offered rescue therapy.

Rescue Medication:

Oral=CQ (3 days, 25mg/kg) together with primaquine (0.25mg/kg/day for 14 days); Intravenous (IV)= Artesunate (4mg/kg/day) for a minimum of 24h and until the patient is able to take oral drug. Then continue with oral DHA-PPQ for 3days.

Radical cure. primaquine treatment will be delayed until the end of the follow up, and given as recommended by the national guidelines, i.e. 0.25mg/kg/day for 14 days to all patients with negative G6PD rapid test.

3.5.3 Follow up From Day 0 until parasite clearance patients will be monitored every 12 hours by blood microscopy at least until Day 3 and longer if necessary until parasite clearance defined as two consecutive negative slides.

At each visit, the patient will be interviewed and examined and a finger prick blood sample will be collected for the following outcomes: two blood slides for LM observation (thick and thin film), 200μl of blood in an EDTA/ACD microtainer tube for DNA extraction, and 2 drops of blood into another microtainer tube containing RNAprotect for RNA extraction. At Day 3, an additional drop of blood will be taken to measure Hb concentration with Hemocue method.

Day 7, 14, 21, 28, 35, 42 Patients will be interviewed and examined, the follow-up form will be completed, and any adverse event documented. A finger prick blood sample will be collected for the following outcomes: two blood slides for LM observation (thick and thin film), 200μl of blood in an EDTA/ACD microtainer tube for DNA extraction, and 2 drops of blood in RNAprotect containing microtainer tube.

In addition, at Day 7, 100μl of blood will be taken on filter paper to determine blood CQ concentration. At Days 7, 14, 28, and 42 Hb concentration (Hemocue) will be measured from finger prick.

Day of P.vivax recurrence: If recurrence is confirmed a further venous blood sample will be collected prior to rescue treatment administration. 100μl of this venous blood will be spotted on filter paper to determine blood CQ concentration, the remaining being used for ex vivo assay and cryopreservation as detailed in Annex VI-C.

3.5.4 Loss to follow-up protocol violations Loss to follow-up occurs when, despite all reasonable efforts, an enrolled patient does not attend the scheduled visits and cannot be found. No treatment outcome will be assigned to these patients. These patients will be classified as lost to follow-up and censored or excluded from the analysis.

Study patients who meet any of the following criteria will be classified as withdrawn: i) withdrawal of consent; ii) failure to complete treatment; iii) serious adverse events necessitating termination of treatment before the full course is completed; iv) enrolment violation; v) voluntary protocol violation; vi) involuntary protocol violation

3.5.5 Laboratory procedures and evaluation Microscopy Three slides (thin/thick blood smears) should be obtained at screening, one being stained rapidly (10% Giemsa for 10 min) for examination in a limited number of fields to ensure the presence of P.vivax asexual forms at a minimum parasitaemia of 250/ul. Once the patient is enrolled, the other two slides will be stained more carefully (3% Giemsa for 45 min). Density, will be expressed as the number of asexual parasites per µl of blood, and calculated dividing the number of asexual parasites by the number of WBCs counted and corrected by the estimated WBCs density (typically 8000 per µl). When the asexual parasite count is less than 10 per 200 WBCs, counting will be done against at least 500 WBCs. A blood slide will be considered negative when examination of 1000 WBCs reveals no asexual parasites.

* Ring stage parasitaemia: The number of ring stages will be counted in all positive slides at Day 0 and at Day of recurrence against 200 asexual parasites; only isolates for which the proportion of ring stages exceeds 65% will be used for the ex vivo drug assay.
* Gametocytes: density will be computed by counting the number of gametocytes per 500 WBCs.

Haemoglobin levels Hb levels will be measured on whole blood collected into micro-cuvette using Hemocue following manufacturer instructions.

Measurement of CQ concentration at Day 7 and day of recurrence from 100 µl of blood expelled onto chromatography paper (31ETCHR, Whatman) Parasite molecular detection and genotyping DNA will be extracted at ITM/NIMPE from finger-prick blood samples collected in microtainers. Molecular confirmation of Plasmodium species at Day 0 will be performed by qPCR targeting 18S ribosomal gene. The same qPCR method will be used to identify and quantify P. vivax infections at Day 0 and follow up samples.

P. vivax genotypes will be identified through PCR amplification of 3 markers particularly effective for finger-printing in clinical trials (MS16, Pv3.2 and msp1F3) followed by capillary gel electrophoresis.

RNA extraction and RT-qPCR for gametocytes RNA will be extracted from RNAprotect samples at ITM/NIMPE using affinity columns and DNAse digestion of genomic DNA. To detect and quantify P. vivax gametocyte stages a reverse transcription qPCR (RT-qPCR) targeting Pvs25 gene transcripts will be done on D0 and in all follow-up samples.

Drug resistance laboratory analysis (Day 0 and of recurrence) Briefly, blood will be centrifuged and plasma will be stored at -20ºC. The upper part of buffy coat will be removed carefully and stored at -20ºC. Red blood cells (RBCs) will be resuspended in PBS (1:1) and leukocytes will be depleted using cellulose columns (Sigma). Filtered cells will be washed and pellet measured before resuspending at 50% hematocrite in McCoy medium (blood medium mixture, BMM, 4ml).

Ex vivo drug sensitivity assays: Briefly, plates with predosed 7-point 2-fold dilutions of CQ, PPQ, DHA and quinine will be prepared following WWARN procedures [http://www.wwarn.org/sites/default/files/INV08_PFalciparumDrugSensitivity.pdf]. Minimal inhibitory concentrations and IC50 will be calculated using the In Vitro Analysis and Reporting Tool (IVART) developed online by the WWARN.

G6PD deficiency test: all patients will be tested for G6PD deficiency using the point-of-care test by CareStart (Access Bio, New Jersey, USA) before PQ treatment.

4. Quality Assurance Site monitoring visits will be scheduled on a regular basis. During these visits, information recorded on the case report forms will be verified against source documents. After the case report forms are collated at the end of the trial, they will be reviewed for completeness and accuracy. The data will be double entered into an electronic database, where specially designed computer checks are used to identify selected protocol violations and data errors.

All blood films on admission will be read at the study site as well as by a senior microscopist at a coordinating centre. In addition, an external quality control will be done at ITM on 10% of randomly selected slides. For each of the molecular assays (qPCR, RT-qPCR and parasite genotyping) 10% of the samples processed at NIMPE will be randomly chosen to be re-analysed at ITM. External quality control of ex vivo drug assay results will be done at ITM where the slides will be re-examined for 10% of randomly chosen isolates.

5. Statistical Analytical Plan The analysis of the Day 42 cure rate will be performed both for the intention-to-treat (ITT) patient population and the evaluable patient population (Per Protocol). Data analyses will be performed using STATA 12 software. For categorical variables percentages and corresponding 95% confidence intervals will be calculated following the Wilson's method. Proportions will be compared by calculating the *2 with Yates' correction or by Fisher's exact test where appropriate. Normally distributed continuous data will be compared by Student's t test and analysis of variance. Data not conforming to a normal distribution will be compared by the Mann-Whitney U test or Kruskal-Wallis analysis of variance. The correlation between 2 continuous variables will be assessed using either the Pearson or Spearman's rank correlation coefficient as required.

The overall risk of treatment failure by Day 28 and by Day 42 will be calculated by Kaplan Meier method, and comparisons between risk groups will be done using the log rank test. The PCR adjusted risk at Day 28 and 42 will also be calculated following the genotyping results of each recurrent P.vivax infection. Parasite clearance time and rate will be estimated using the PCE online tool developed by WWARN (http://www.wwarn.org/toolkit/data-management/parasite-clearance-estimator). The Mean IC50 and IC90 for CQ will be estimated using the In vitro Analysis and reporting tool (IVART) developed by WWARN (http://www.wwarn.org/toolkit/data-management/ivart).

Hematological changes will be evaluated by measuring the changes in Hb concentration between day0, 3, 7, 14, 28 and 42, respectively.

6. Ethical Issues 6.1 Ethical clearance to conduct the study will have been obtained from the Ethics Committee of the NIMPE, Hanoi and from the Ethics Committee of the University of Antwerp, as well as from the Institutional Review Board at the ITM, Anwerp.

6.2 Consent Process Patients will be included in the study only if they (or parents or guardians of children) give informed consent. The consent request is available in English and translated into Vietnamese to be read entirely to the patient, parent or guardian. Details about the trial and its benefits and potential risks will be explained. Once any questions have been answered, a signature will be requested on the document. If the patient is illiterate, a literate witness must sign; if possible, the signatory will be selected by the participant and will have no connection to the research team.

ELIGIBILITY:
Inclusion Criteria:

* Mono-infection of P. vivax by light microscopy (LM) with asexual parasite density >250/µl
* Age ≥1year
* Axillary temperature ≥ 37.5º C and/or history of fever during the previous 48 hours;
* Patient or caregiver consent to enrolment and agree to sampling and return visits;

Exclusion Criteria:

* General danger signs or symptoms of severe malaria (as per WHO definitions; Annex I);
* Signs or symptoms of severe malnutrition, defined as weight-for-age ≤ 3 standard deviations below the mean (NCHS/WHO normalized reference values, Annex II);
* Slide confirmed infection with any other Plasmodium species (including mixed infections);
* Severe anaemia, defined as haemoglobin (Hb) <7g/dl in adults and <5g/dl in children;
* Known hypersensitivity to any of the drugs being evaluated;
* Presence of fever due to illness other than malaria;
* History of serious and/or chronic medical condition (cardiac, renal, hepatic diseases, sickle cell disease, HIV/AIDS);
* Pregnancy (confirmed by rapid test) or breastfeeding;
* Regular use of medication that may interfere with antimalarial pharmacokinetics;

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Adequate Clinical and Parasitological Response (ACPR) at day 42 after treatment with Chloroquine. | day 42
  This outcome will be measured at day42 of follow-up. Treatment outcomes such as ACPR, early or late clinical failures are defined following WHO guidelines;

SECONDARY OUTCOMES:
Ex vivo susceptibility of P. vivax isolates to QN, DHA , PPQ and CQ (Mean IC50 and IC90) | At day0 and day of recurrence of P.vivax parasitemia after initial parasite clearance assessed up to day 42
  Individual and mean IC50 and IC90 values will be computed for each drug using the IVART tool available online (http://www.wwarn.org/tools-resources/toolkit/analyse/ivart)

OTHER OUTCOMES:
Number of patients carrying asexual parasites during 42 days follow up | From day0 to day 42
  asexual parasite forms will be detected by qPCR. This outcome will be measured for each sampling time point.
Number of patients with parasites carrying molecular markers of Plasmodium vivax resistance to CHL at day 0 and among recurrent vivax infections | From day 0 to day42
  All parasites at day0 will be genotyped and processed by whole genome sequencing to identify molecular markers of CHL resistance. The same analysis will be done for any P. vivax recurrence occurring during the 42-day follow-up.
The number of patients with glucose-6-phosphate dehydrogenase (G6PD) deficiency measured by rapid test | day 42
  All patients will be tested for G6PD deficiency by a rapid test (CareStart) before given the radical cure treatment with primaquine.
Number of patients carrying sexual parasites during 42 days follow up | From day0 to day 42
  sexual parasite forms will be detected by RT-qPCR. This outcome will be measured for each sampling time point.
Number of patients with allelic variants of glucose-6-phosphate dehydrogenase (G6PD) deficiency | Day 42
  G6PD allelic variants will be assessed by allele-specific qPCR assay

CONTACTS AND LOCATIONS:
Overall Officials: Duong Tran, MD, PhD, Principal Investigator — National Institute of Malariology Parasitology Entomology, Hanoi, Vietnam; Anna Rosanas-Urgell, MD, PhD, Principal Investigator — Institute of Tropical Medicine, Antwerp, Belgium
Locations (1):
- Chu R Cam, Pleiku, Gia Lai, Vietnam

REFERENCES:
- [Background] Rosanas-Urgell A, Mueller D, Betuela I, Barnadas C, Iga J, Zimmerman PA, del Portillo HA, Siba P, Mueller I, Felger I. Comparison of diagnostic methods for the detection and quantification of the four sympatric Plasmodium species in field samples from Papua New Guinea. Malar J. 2010 Dec 14;9:361. doi: 10.1186/1475-2875-9-361. PMID 21156052
- [Background] Koepfli C, Mueller I, Marfurt J, Goroti M, Sie A, Oa O, Genton B, Beck HP, Felger I. Evaluation of Plasmodium vivax genotyping markers for molecular monitoring in clinical trials. J Infect Dis. 2009 Apr 1;199(7):1074-80. doi: 10.1086/597303. PMID 19275476
- [Background] Wampfler R, Mwingira F, Javati S, Robinson L, Betuela I, Siba P, Beck HP, Mueller I, Felger I. Strategies for detection of Plasmodium species gametocytes. PLoS One. 2013 Sep 27;8(9):e76316. doi: 10.1371/journal.pone.0076316. eCollection 2013. PMID 24312682
- [Background] Auburn S, Marfurt J, Maslen G, Campino S, Ruano Rubio V, Manske M, Machunter B, Kenangalem E, Noviyanti R, Trianty L, Sebayang B, Wirjanata G, Sriprawat K, Alcock D, Macinnis B, Miotto O, Clark TG, Russell B, Anstey NM, Nosten F, Kwiatkowski DP, Price RN. Effective preparation of Plasmodium vivax field isolates for high-throughput whole genome sequencing. PLoS One. 2013;8(1):e53160. doi: 10.1371/journal.pone.0053160. Epub 2013 Jan 4. PMID 23308154
- [Background] Kerlin DH, Boyce K, Marfurt J, Simpson JA, Kenangalem E, Cheng Q, Price RN, Gatton ML. An analytical method for assessing stage-specific drug activity in Plasmodium vivax malaria: implications for ex vivo drug susceptibility testing. PLoS Negl Trop Dis. 2012;6(8):e1772. doi: 10.1371/journal.pntd.0001772. Epub 2012 Aug 7. PMID 22880143
- [Background] Borlon C, Russell B, Sriprawat K, Suwanarusk R, Erhart A, Renia L, Nosten F, D'Alessandro U. Cryopreserved Plasmodium vivax and cord blood reticulocytes can be used for invasion and short term culture. Int J Parasitol. 2012 Feb;42(2):155-60. doi: 10.1016/j.ijpara.2011.10.011. Epub 2011 Dec 27. PMID 22240310
- [Background] Kim S, Nguon C, Guillard B, Duong S, Chy S, Sum S, Nhem S, Bouchier C, Tichit M, Christophel E, Taylor WR, Baird JK, Menard D. Performance of the CareStart G6PD deficiency screening test, a point-of-care diagnostic for primaquine therapy screening. PLoS One. 2011;6(12):e28357. doi: 10.1371/journal.pone.0028357. Epub 2011 Dec 2. PMID 22164279
- [Derived] Rovira-Vallbona E, Van Hong N, Kattenberg JH, Huan RM, Binh NTH, Ngoc NTH, Guetens P, Hieu NL, Hien NTT, Sang VT, Long ND, Sauve E, Duong TT, Xa NX, Erhart A, Rosanas-Urgell A. High Proportion of Genome-Wide Homology and Increased Pretreatment pvcrt Levels in Plasmodium vivax Late Recurrences: a Chloroquine Therapeutic Efficacy Study. Antimicrob Agents Chemother. 2021 Jul 16;65(8):e0009521. doi: 10.1128/AAC.00095-21. Epub 2021 Jul 16. PMID 34031050